CLINICAL TRIAL: NCT00245596
Title: An Open Label, Multicenter Study to Measure Treatment Responsiveness of Quality of Sexual Life Questionnaire in the Female Partner of Men With Erectile Dysfunction Treated With Viagra (Sildenafil Citrate)
Brief Title: Evaluation of the Index of Sexual Life Questionnaire
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481210
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
The purpose of the study is to assess the sensibility of the ISL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

ED patient must:

* Be male, 18 years of age with no upper age limit;
* Have a documented clinical diagnosis of erectile dysfunction confirmed by an Erectile Function (IIEF) score 25. Erectile dysfunction is defined as "the inability to achieve and/or maintain an erection of the penis sufficient to permit satisfactory sexual performance" (Impotence-NIH Consensus Conference, JAMA 1993, 270: 83-90);
* Have a stable female partner for at least 6 months prior to screening.

Exclusion Criteria:

* Have a known hypersensitivity to sildenafil or any component of the study medication; medical history of treatment-related intolerable side effects to sildenafil
* Be currently prescribed, taking and/or likely to be treated with nitrates or nitric oxide donors in any form on either a regular or intermittent basis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-10

PRIMARY OUTCOMES:
Treatment responsiveness of a new quality of sexual life questionnaire for female partners of men with erectile dysfunction.

SECONDARY OUTCOMES:
The correlation between ED patients' partner quality of sexual life changes and patient's efficacy measures and these changes and patient reported outcomes of self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- France (9):
  - Pfizer Investigational Site, Amphion-les-Bains
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, La Rochelle
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Émilion
  - Pfizer Investigational Site, Thionville
  - Pfizer Investigational Site, Toulouse

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481210&StudyName=Evaluation+of+the+Index+of+Sexual+Life+Questionnaire